CLINICAL TRIAL: NCT05864066
Title: The Role of Cyclin-dependent Kinase Inhibitor 2A (P16 INK4a) (Placental Senescence Marker) on Labor-related Signals Through Progesterone Receptors Expression in Human Placenta
Brief Title: Cyclin-dependent Kinase Inhibitor 2A (Placental Senescence Marker) on Labor-related Signals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma El-sayed Moustafa, principal investigator, Assiut University
Other Study IDs: P16 INK4a and PR
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Women in preterm delivery with GA < 36 weeks.
- 2: Women not in labor undergoing elective C-section with GA between 36 and 40 weeks.
- 3: Women following spontaneous labor (without being induced) with GA between 36 and 40 weeks.

SUMMARY:
Onset of labor in human is initiated by progesterone withdrawal. Over many decades researchers had proposed hypotheses to explain the functional withdrawal of progesterone. These hypotheses were through the sequestration of active progesterone by corticosteroid-binding globulin, a decrease in active progesterone metabolite levels and changes in the ratio of progesterone receptor (PR) isoforms (nuclear progesterone receptors A (nPRA) and nuclear progesterone receptors B (nPRB)). Progesterone performs its action non-genomically through binding to membrane receptors and genomically via binding to nPRs. PRA is the less active or inactive form of progesterone receptors and shorter in amino acid sequence than PRB, the active form of the receptors.

DETAILED DESCRIPTION:
Another mechanism was done through transcriptional co-activators, repressors inflammation resulting in nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kB) mediated PR suppression. Previous study had explored that the uterine myometrium as the site of this functional withdrawal. There is also a clock that can determine the length of human pregnancy resides in the placenta and functional progesterone withdrawal likely occurs in this organ as well.

Ageing is a process that causes deterioration in function at the cellular, tissue and organ levels. Telomeres are protective caps made of nucleoprotein molecules located at the end of chromosomes and are necessary for protection against breaks at DNA ends, fusion of chromosome ends and chromosome degradation.

Telomeres are shortened with each cell division. The rate at which this occurs is accelerated by certain stressors such as oxidative stress. When telomeres reach a dangerously short length the process of cellular senescence initiates through which cells irreversibly stop growing and dividing by arresting their cell cycle and gradually ageing (becoming senescent).

Cellular senescence is a state of irreversible cell cycle arrest resulting from high levels of P16 INK4a as well as tumour 15 suppressors p53 and retinoblastoma tumour suppressor protein. Senescent cells markedly have an ability to change gene expression patterns with overexpression of anti-apoptotic Bcl-2 leading to resistance to apoptosis and in parallel increase NFκB activity results in the expression of proinflammatory cytokines and chemokines. As pregnancy comes to term, decidual cells show many features of senescence including secretion of senescence-associated secretory phenotype (SASP) factors such as interleukin-6 (IL-6). A gradual process of decidual senescence may be critical for driving the cellular and tissue changes that contribute to labor onset at term. If ageing of the placenta normally determines pregnancy duration, this means that premature placental ageing will lead to preterm labor onset.

According to World Health Organization (WHO), the American Academy of Pediatrics (AAP), and the American College of Obstetricians and Gynecologists (ACOG), preterm birth is defend as babies born alive before 37 weeks of pregnancy are completed. Each year, 15million babies are born preterm in the world. The National Center for Health Statistics of the Centers for Disease Control and Prevention generally reports data on three categories of preterm birth: overall preterm (< 37 weeks 'gestation), moderately preterm (between 32 and 36 weeks' gestation) and very preterm births (< 32 weeks' gestation). Late preterm infants are born at a gestational age between 34 weeks and less than37 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who will come for termination of pregnancy by caesarean section or vaginal delivery.
* Gestational age is between 28 to < 37 weeks for preterm labor and 37 to 40 weeks for term labor.
* The age range of women is between18- 40 years.

Exclusion Criteria:

* Acute or chronic infectious diseases or other chronic illness
* Autoimmune diseases
* PE complicated with Eclampsia, DIC or HELP syndrome
* Congenital anomaly of the uterus
* History of trauma
* Twins pregnancy
* Congenital anomalies of the fetus
* Fetal growth restriction

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women who will come for termination of pregnancy
Sampling Method: Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
P16 INK4a | one year
  1.Evaluating the role of cyclin-dependent kinase inhibitor 2A (P16 INK4a) placental senescence marker to predict time of labor.

SECONDARY OUTCOMES:
PR | one year
  2.Local effect of cyclin-dependent kinase inhibitor 2A (P16 INK4a) placental senescence marker on progesterone receptors expression in human placenta.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Grazul-Bilska AT, Thammasiri J, Kraisoon A, Reyaz A, Bass CS, Kaminski SL, Navanukraw C, Redmer DA. Expression of progesterone receptor protein in the ovine uterus during the estrous cycle: Effects of nutrition, arginine and FSH. Theriogenology. 2018 Mar 1;108:7-15. doi: 10.1016/j.theriogenology.2017.11.008. Epub 2017 Nov 20. PMID 29175682
- [Background] Jacobsen BM, Horwitz KB. Progesterone receptors, their isoforms and progesterone regulated transcription. Mol Cell Endocrinol. 2012 Jun 24;357(1-2):18-29. doi: 10.1016/j.mce.2011.09.016. Epub 2011 Sep 17. PMID 21952082
- [Background] Kidus F, Woldemichael K, Hiko D. Predictors of neonatal mortality in Assosa zone, Western Ethiopia: a matched case control study. BMC Pregnancy Childbirth. 2019 Mar 29;19(1):108. doi: 10.1186/s12884-019-2243-5. PMID 30925903
- [Background] Kowalik MK, Rekawiecki R, Kotwica J. Expression of membrane progestin receptors (mPRs) in the bovine corpus luteum during the estrous cycle and first trimester of pregnancy. Domest Anim Endocrinol. 2018 Apr;63:69-76. doi: 10.1016/j.domaniend.2017.12.004. Epub 2018 Jan 11. PMID 29413904
- [Background] Kumari R, Jat P. Mechanisms of Cellular Senescence: Cell Cycle Arrest and Senescence Associated Secretory Phenotype. Front Cell Dev Biol. 2021 Mar 29;9:645593. doi: 10.3389/fcell.2021.645593. eCollection 2021. PMID 33855023
- [Background] Martin JA, Hamilton BE, Osterman MJK, Driscoll AK. Births: Final Data for 2018. Natl Vital Stat Rep. 2019 Nov;68(13):1-47. PMID 32501202
- [Background] Menon R, Bonney EA, Condon J, Mesiano S, Taylor RN. Novel concepts on pregnancy clocks and alarms: redundancy and synergy in human parturition. Hum Reprod Update. 2016 Sep;22(5):535-60. doi: 10.1093/humupd/dmw022. Epub 2016 Jun 30. PMID 27363410